CLINICAL TRIAL: NCT01759563
Title: Safety and Feasibility Study of Nasopharyngeal Cooling (RhinoChill Device) During Transcutaneous Aortic Valve Implantation
Brief Title: Oxygenation of the Cerebrum and Cooling During TAVI - Part I
Acronym: OCCTAVI-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Prof Dr Cathy De Deyne, Prof Dr Jo Dens, Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OCCTAVI-I; COBRA Research Group (Other: Cardio+Brain Research Group UHasselt)
Record Dates: First submitted 2012-12-27; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: TAVI; Targeted Brain Cooling; Neuroprotection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm study (Other)
  Interventions: Device: nasopharyngeal targeted brain cooling

INTERVENTIONS:
Device: nasopharyngeal targeted brain cooling
  Other Names: RhinoChill Device, BeneChill company

SUMMARY:
Assessment of safety and feasibility of using a nasopharyngeal cooling technique to provide targeted brain cooling during percutaneous implantation of aortic valves. Was it possible to obtain brain temperatures below 34° within a reasonable time interval (max of 1hr) without delaying the procedure of valve implantation.

DETAILED DESCRIPTION:
OCCTAVI-I Protocol

6 patients selected for Transcutaneous Aortic Valve Implantation (TAVI)-procedure will be subjected to intra-operative transnasal cooling (RhinoChill) ; cooling will be started after induction of anesthesia until tympanic temperature achieves 34° (cooling will be continued until 33°C of tympanic temperature, below 33°C active cooling will be stopped)

No intra-aortic catheter will be inserted before tympanic temperature reaches 34°

The aim of this study is to test the safety (as referring to routinely used neuromonitoring : ForeSight cerebral tissue oxygen saturation (SctO2) monitoring; and as referring to cardiovascular stability : blood pressure & heartrate) and feasibility (as referring to temperature characteristics) of brain cooling during TAVI (cerebral (or tympanic) cooling rate, differential tympanic-rectal cooling rate, rectal cooling rate, time needed to obtain tympanic temperature below 34°)

Patients will be monitored with FORE-SIGHT cerebral oximeter (regional cerebral oxygen saturation, sensors placed on patient's forehead) and BIS VISTA (bilateral continuousEEG).

Tympanic temperature will be measured every 5 minutes while oesophageal and blood temperature will be continuously measured.

* Neuromonitoring (Fore-Sight, Bispectral Index (BIS) Vista) will be started before induction of anesthesia and cooling
* Transnasal cooling will be started after induction of anesthesia until a target tympanic temperature of 34°C
* Core temperature will not be monitored by esophageal (caveat interaction TEE probe), but by rectal and blood temperature
* TAVI-procedure will be started at a tympanic temperature of 34°C
* Arterial CO2 tension (PaCO2) will be checked every 30 minutes intra-operatively (target=normocapnia) by arterial blood gas analysis to maintain strict normocapnia
* and the end of the TAVI-procedure, patient will be rewarmed at a max rate of 0.8°/h by total body bair hugger
* when patient reaches tympanic and systemic (rectal) temperature of 35.5°C, extubation can be performed

ELIGIBILITY:
Inclusion Criteria:

* pts eligible for TAVI interventions

Exclusion Criteria:

* urgent intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome is the brain temperature obtained after initiation of nasopharyngeal cooling. Safety-outcome includes local or systemic side-effects of used cooling technique. | Day1: start of cooling until brain temperature above 35.5°C
  By the use of nasopharyngeal cooling, brain temperature will be decreased. Time to brain temperature below 34° will be recorded. Local side effects could occur due to the use of this specific nasopharyngeal cooling technique and systemic side effects (especially cardiovascular) could occur due to the initiation of hypothermia

SECONDARY OUTCOMES:
changes in cerebral oxygenation (NIRS Fore-Sight technology) induced by targeted brain cooling | Day 1: start of cooling until brain temperature above 35.5°C
  NIRS (or Near-infrared Spectroscopy) enables non-invasive monitoring of cerebral oxygen saturation during TAVI procedure and during the installation of targeted brain cooling. NIRS will be used as cerebral monitoring technique during this study protocol

OTHER OUTCOMES:
Influence of targeted brain cooling on systemic core temperature | Day 1: start of cooling until brain temperature above 35.5°C
  Induction of nasopharyngeal cooling and targeted brain cooling will result in systemic hypothermia. Systemic temperature (rectal temperature) will be recorded to assess the influence of nasopharyngeal cooling on systemic body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Cathy De Deyne, Md, PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

REFERENCES:
- [Background] Castren M, Nordberg P, Svensson L, Taccone F, Vincent JL, Desruelles D, Eichwede F, Mols P, Schwab T, Vergnion M, Storm C, Pesenti A, Pachl J, Guerisse F, Elste T, Roessler M, Fritz H, Durnez P, Busch HJ, Inderbitzen B, Barbut D. Intra-arrest transnasal evaporative cooling: a randomized, prehospital, multicenter study (PRINCE: Pre-ROSC IntraNasal Cooling Effectiveness). Circulation. 2010 Aug 17;122(7):729-36. doi: 10.1161/CIRCULATIONAHA.109.931691. Epub 2010 Aug 2. PMID 20679548